CLINICAL TRIAL: NCT03434964
Title: Preliminary Evaluation of the AIFib Software in Real Time as a Medical Decision Aid for the Detection of Atrial Fibrillation Driver
Brief Title: Ev-AIFIB Preliminary Evaluation of the AIFib Software
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Other Study IDs: HSJ_EvAIFIB_2018
Record Dates: First submitted 2018-02-07; First posted 2018-02-15 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2020-04

CONDITIONS: Software Performance Evaluation a Posteriori

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the intraoperative effectiveness of the AIFIB software in real time in the detection of atrial fibrillation drivers during an ablation procedure. — Real-time validation by an expert operator of the correct detection of atrial fibrillation driver

SUMMARY:
To evaluate the intraoperative effectiveness of the AIFIB software in real time in the detection of atrial fibrillation drivers during an ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Etiology in the following list:
* Atrial fibrillation for which a conventional anatomical approach alone (pulmonary vein isolation) is not performed: persistent AF, long standing persistent AF paroxysmal AF (redo), paroxysmal AF
* Atrial tachycardia de novo or secondary to AF ablation.

Exclusion Criteria:

* Contraindication to AF ablation
* Major bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years with an indication of ablation of FA or TA
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Software performance evaluation a posteriori | during the ablation procedure
  real-time validation by the second operator of the correct detection of atrial fibrillation driver

SECONDARY OUTCOMES:
Indirect evaluation of the clinical effectiveness of the software | during the ablation procedure
  AF stopping rate by removal of the areas detected by the main operator and the software

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Groupe Hopitaux Institut Catholique de Lille, Lille
  - Clinique de l'Infirmerie Protestante, Lyon
  - Saint Joseph Hospital, Marseille
  - Clinique Ambroise Paré, Neuilly, Neuilly-sur-Seine
  - CHU NICE Pasteur, Nice
  - IHCPS Massy, Paris
  - Centre de cardiologie du Nord, Saint-Denis
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No